CLINICAL TRIAL: NCT04125095
Title: Estimating Setup Uncertainty in Pediatric Proton Therapy Using Volumetric Images
Status: Active, not recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SJPROTON2
Record Dates: First submitted 2019-10-10; First posted 2019-10-14 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Cancer
Keywords: Proton therapy, Children and adolescents, Image guidance, Setup uncertainty
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Head Scans: Includes patients receiving proton therapy for tumors in the brain, skull, and head and neck region. The same patient could potentially contribute to both cohorts if he/she receives radiation to both head and body sites.
- Body Scans: Includes proton irradiation to shoulders, thorax, abdomen, pelvis, spine (thoracic or lumbar), extremities, and other body sites. The same patient could potentially contribute to both cohorts if he/she receives radiation to both head and body sites.

SUMMARY:
This research study establishes a repository for imaging data generated during image-guided proton therapy for various pediatric cancers. The data facilitate the estimation of patient positioning uncertainty, the comparison of image guidance methods, and the identification of factors contributing to large setup deviations to improve the accuracy of radiation therapy in the future.

Primary Objective

To establish a repository of imaging data acquired during the radiation therapy course with linked radiation treatment plans and clinical information from pediatric patients of all cancer types receiving image-guided proton therapy to facilitate secondary and exploratory objectives.

Secondary Objectives

* To estimate distributions of patient setup uncertainty measured with daily pre- treatment volumetric cone beam computed tomography (CBCT) scans.
* To compare patient setup corrections derived based on 2D (orthogonal radiographs) and 3D (volumetric CBCT scans) image guidance.
* To assess residual setup errors after CBCT-guided correction based on post- correction repeat CBCT.
* To estimate distributions and time trends of patient motion during a radiation therapy course based on weekly pre- and post-treatment CBCT scans.
* To identify clinical and treatment factors that contribute to significantly large setup uncertainty and intra-fractional movement in pediatric patients.

Exploratory Objectives

* To determine variation in patient anatomy using images acquired during the treatment course.
* To evaluate the usefulness of on-treatment CBCT scans for detecting daily changes in proton ranges, evaluating deviations from planned tumor dosimetry, and triggering adaptive replanning.

DETAILED DESCRIPTION:
Image guidance data collected in this study include daily volumetric pre-treatment CBCT for image guidance, post-correction CBCT, weekly post-treatment CBCT, and 2D orthogonal radiographs. Setup uncertainty will be estimated for head and body cohorts separately, further divided into different anatomic sites. The usefulness and necessity of daily volumetric image guidance for pediatric proton therapy patients will be determined. Knowledge gained from this study will provide a basis for reducing patient positioning uncertainty and designing optimal treatment plans for pediatric patients receiving proton therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient will receive proton therapy of ≥5 daily fractions.
* Research participant or legal guardian/representative gives written informed consent.

Exclusion Criteria:

* Unwillingness of research participant or legal guardian/representative to give written informed consent.
* If patients previously enrolled in this study and completed protocol-specified imaging scans but return for re-irradiation, they will not be eligible to participate again.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric patients of all cancer types who undergo at least 5 daily treatments of proton therapy.
Sampling Method: Non-Probability Sample
Enrollment: 367 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Site-specific distributions of patient setup uncertainty. | 5 years after activation
  The numbers of subjects enrolled in the head cohort and the body cohort.

SECONDARY OUTCOMES:
Differences in setup errors calculated from orthogonal radiographs and cone beam computed tomography (CBCT) | 5 years
  This is to determine if setup corrections estimated from orthogonal radiographs are similar to those from volumetric imaging. The differences of each positional shift (x, y, z, pitch, roll, yaw) are measured.
Residual errors after image-guided setup corrections | 5 years
  This is to determine if residual setup errors are submillimeter after image guidance with robotic cone beam computed tomography and 6 degree-of-freedom patient positioner. Residual errors differences for six parameters (x, y, z, pitch, roll, yaw) are measured.
Distributions of intra-fractional patient motion | 5 years
  This is to estimate the change in patient position during a treatment fraction based on pre- and post-fractional volumetric imaging. The differences of each positional shift (x, y, z, pitch, roll, yaw) are measured.
Risk factors of large setup uncertainty and intra-fractional movement | 5 years
  Risk factors (e.g., age, anesthesia, and anatomic site) that associate with the significantly large setup uncertainty and intra-fractional movement will be identified. The association with p value between age and setup uncertainty is measured.
Risk factors of large setup uncertainty and intra-fractional movement | 5 years
  Risk factors (e.g., age, anesthesia, and anatomic site) that associate with the significantly large setup uncertainty and intra-fractional movement will be identified. The association with p value between anesthesia and setup uncertainty is measured.
Risk factors of large setup uncertainty and intra-fractional movement | 5 years
  Risk factors (e.g., age, anesthesia, and anatomic site) that associate with the significantly large setup uncertainty and intra-fractional movement will be identified. The association with p value between anatomic site and setup uncertainty is measured.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-ho Hua, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Background] Becksfort J, Uh J, Saunders A, Byrd JA, Worrall HM, Marker M, Melendez-Suchi C, Li Y, Chang J, Raghavan K, Merchant TE, Hua CH. Setup Uncertainty of Pediatric Brain Tumor Patients Receiving Proton Therapy: A Prospective Study. Cancers (Basel). 2023 Nov 20;15(22):5486. doi: 10.3390/cancers15225486. PMID 38001746
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

DOCUMENTS (1):
  • Informed Consent Form (2021-09-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT04125095/ICF_000.pdf